CLINICAL TRIAL: NCT00262860
Title: Phase II Pilot Study of Bortezomib (VELCADE®) and Gemcitabine for Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: Bortezomib and Gemcitabine Hydrochloride in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jonathan Friedberg, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000448635; URCC-U9404; URCC-RSRB-10368; MILLENNIUM-VEL-03-079; LILLY-B9E-US-X433; DFCI-04388
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-03

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bortezomib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib, Gemcitabine Hdrochloride (Experimental)
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bortezomib
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with gemcitabine hydrochloride may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with gemcitabine hydrochloride works in treating patients with relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate (partial and complete response) in patients with relapsed or refractory Hodgkin's lymphoma treated with bortezomib and gemcitabine hydrochloride.

Secondary

* Determine the safety and toxic effects of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.
* Correlate NF-kB inhibition and proteasome activity with response in patients treated with this regimen.

OUTLINE: This is a multicenter, pilot study.

Patients receive bortezomib IV on days 1, 4, 8, and 11 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma

  * Recurrent or refractory disease after prior standard combination chemotherapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 1 cm by physical exam or imaging studies
* No history of non-Hodgkin's lymphoma
* No history of other hematological malignancy

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN) (unless due to Gilbert's disease or involvement by Hodgkin's lymphoma)
* AST ≤ 3 times ULN (unless due to involvement by Hodgkin's lymphoma)

Renal

* Creatinine clearance ≥ 30 mL/min

Cardiovascular

* Ejection fraction ≥ 40% by MUGA or echocardiogram (in patients with a history of cardiac disease)

Pulmonary

* Must not require supplemental oxygen therapy

Immunologic

* No known HIV infection
* No uncontrolled bacterial, viral, or fungal infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy requiring therapy
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No hypersensitivity to boron
* No hypersensitivity to mannitol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 30 days since prior monoclonal antibody therapy for Hodgkin's lymphoma
* More than 6 months since prior autologous stem cell transplantation
* No prior allogeneic stem cell transplantation
* No concurrent sargramostim (GM-CSF)
* No concurrent pegfilgrastim or filgrastim (G-CSF)
* No concurrent interleukin-11(oprelvekin)

Chemotherapy

* See Disease Characteristics
* More than 30 days since prior chemotherapy for Hodgkin's lymphoma
* No prior treatment with gemcitabine hydrochloride

Endocrine therapy

* More than 30 days since prior corticosteroid therapy for Hodgkin's lymphoma
* No concurrent corticosteroid therapy

Radiotherapy

* More than 30 days since prior radiotherapy for Hodgkin's lymphoma

Other

* No prior treatment with bortezomib
* More than 14 days since prior investigational drugs
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Friedberg, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Result] Mendler JH, Kelly J, Voci S, Marquis D, Rich L, Rossi RM, Bernstein SH, Jordan CT, Liesveld J, Fisher RI, Friedberg JW. Bortezomib and gemcitabine in relapsed or refractory Hodgkin's lymphoma. Ann Oncol. 2008 Oct;19(10):1759-64. doi: 10.1093/annonc/mdn365. Epub 2008 May 25. PMID 18504251

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib, Gemcitabine Hydrochloride: bortezomib
  gemcitabine hydrochloride
  Bortezomib was administered at a dose of 1 mg/m2 on days 1, 4, 8,and 11 of a 21-day schedule. Gemcitabine was administered at a dose of 800 mg/m2 on days 1 and 8 of the same 21-day schedule.
Period: Overall Study
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Started | 18
Completed | 16
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 36 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16
  Black | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate After 2 Courses of Therapy
Description: Response was evaluated after two cycles of therapy using the 1999 Cheson response criteria. All responses were based on CT scans. The criteria that were developed include anatomic definitions of response, with normal lymph node size after treatment of 1.5 cm in the longest transverse diameter by computer-assisted tomography scan. A designation of complete response/unconfirmed was adopted to include patients with a greater than 75% reduction in tumor size after therapy but with a residual mass, to include patients-especially those with large-cell NHL-who may not have residual disease. For patients who had FDG-PET imaging, metabolic response was defined as a decrease in the standardized uptake value in target lesions (regions of abnormal FDG uptake on pretreatment FDG-PET images) to below three on posttreatment FDG-PET imaging). All PET scans were reviewed and interpreted by a single radiologist (SV).
Time Frame: 21 Days/course for up to 2 courses
Measure: Number; unit: participants
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Number analyzed (Participants) | 18
participants | 4

2. Secondary Outcome: Change in Proteasome Activity Compared to Baseline (Cycle 1)
Description: Peripheral blood (40 ml) was collected on cycle 1, day 1 of prebortezomib at baseline and 2 hrs post-bortezomib treatment. The samples were refrigerated at 4C and processed within 36 h of collection. Frozen cell lysates were thawed and the proteasome activity in 10 microliters was determined using a spectroflourometric 20S proteasome assay kit. Samples were run in triplicate on two separate days. The percent change between baseline and 2 hrs (day1, cycle 1) was calculated.
Time Frame: baseline to 2 hours
Population: Samples were not collected on one patient, so only 17 patients were analyzed.
Measure: Median (Full Range); unit: Percentage of change in proteosome activ
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Number analyzed (Participants) | 17
Percentage of change in proteosome activ | -50 [-77 to 39]

3. Secondary Outcome: Change in Proteasome Activity Compared to Baseline (Cycle 2)
Description: Peripheral blood (40 ml) was collected at baseline and 1-2 weeks after cycle 2, day 11 post-bortezomib treatment. The samples were refrigerated at 4C and processed within 36 h of collection. Frozen cell lysates were thawed and the proteasome activity in 10 microliters was determined using a spectroflourometric 20S proteasome assay kit. Samples were run in triplicate on two separate days. The percent change between baseline and 2 hrs (day1, cycle 1) was calculated.
Time Frame: baseline and 1-2 weeks after cycle 2, day 11
Population: Samples were not collected on one patient, so only 17 patients were analyzed.
Measure: Median (Full Range); unit: percentage of change in proteosome activ
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Number analyzed (Participants) | 17
percentage of change in proteosome activ | -57 [-92 to 223]

ADVERSE EVENTS:
Time Frame: days 1 and 8 of each cycle of therapy, up to 2 months
Arm/Group | Bortezomib, Gemcitabine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib, Gemcitabine Hydrochloride (N=18)
neutropenia (Blood and lymphatic system disorders) | 5
leukopenia (Blood and lymphatic system disorders) | 3
thrombocytompenia (Blood and lymphatic system disorders) | 2
elevated transaminases (Hepatobiliary disorders) | 3
hyperglycemia (Vascular disorders) | 1
abdominal pain/cramps (General disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 1
headache/migraine (Nervous system disorders) | 1
sepsis (Infections and infestations) | 1
DVT near line (Vascular disorders) | 1
worsening leg ulcer (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib, Gemcitabine Hydrochloride (N=18)
neutropenia (Blood and lymphatic system disorders) | 5
leukopenia (Blood and lymphatic system disorders) | 7
thrombocytopenia (Blood and lymphatic system disorders) | 8
elevated transaminases (Hepatobiliary disorders) | 4
hyperglycemia (Endocrine disorders) | 3
abdominal pain/cramps (Gastrointestinal disorders) | 2
anemia (Blood and lymphatic system disorders) | 8
pain (General disorders) | 7
hypocalcemia (Blood and lymphatic system disorders) | 6

LIMITATIONS AND CAVEATS:
Trial was stopped early by the Data Safety Monitoring Committee due to unexpected toxicity with no improvement in the response rate compared with gemcitabine alone. Trial was prespecified to be stopped early if these criteria were met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes